CLINICAL TRIAL: NCT04224831
Title: Treatment of Chronic Recalcitrant or Unresponsive Central Serous Chorioretinopathy Via Electromagnetic Stimulation And Platelet- Rich Plasma
Brief Title: Treatment of Chronic Central Serous Chorioretinopathy Via Electromagnetic Stimulation and Platelet- Rich Plasma
Acronym: CSCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Universitesi Teknokent (Other)
Responsible Party: Principal Investigator, Umut Arslan, Principle investigator, MD, Ankara Universitesi Teknokent
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03.10.2018/02
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Central Serous Chorioretinopathy; Chronic Central Serous Chorioretinopathy
Keywords: Central serous chorioretinopathy; Electromagnetic stimulation; Platelet rich plasma; Growth factors; Iontophoresis
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Iontophoresis

STUDY DESIGN:
Intervention Model Description: Prospective, open label study; The cases resistant to all known conventional treatment methods were compared before and after the application. The control group cannot be formed because there are cases resistant to all treatment methods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before application (Active Comparator): The chronic CSCR cases included here meet one or more of the following criteria:
  * Complaints of recurrent symptoms lasting longer than 3 months;
  * Recalcitrant or unresponsive to all known current treatment modalities including PDT and MPL;
  * Typical B-scan SD-OCT findings of chronicity such as elongation of photoreceptor outer segments indicating chronic nature of sub-macular fluid and/or the presence of serous flat-irregular RPED and focal areas of thickened RPE that lie below the collection of SRF;
  * Widespread RPE/photoreceptor damage, RPE mottling and atrophy along with chronic submacular fluid;
  * Widespread multifocal areas of chronic serous retinal detachment and/or flat-irregular RPEDs in those eyes that effective and reliable laser application is impossible.
  Interventions: Combination Product: Source of growth factors: autologous platelet-rich plasma (aPRP) + repetitive electromagnetic stimulation for iontophoresis
- After application (Active Comparator): The changes in SMT, CMT, DRCD, and BCVA before and after the interventions were compared.
  Interventions: Combination Product: Source of growth factors: autologous platelet-rich plasma (aPRP) + repetitive electromagnetic stimulation for iontophoresis

INTERVENTIONS:
Combination Product: Source of growth factors: autologous platelet-rich plasma (aPRP) + repetitive electromagnetic stimulation for iontophoresis — Autologous platelet rich plasma is containing many types of growth factors (GFs) such as epithelial growth factor (EGF), fibroblast growth factor (FGF), transforming growth factor (TGF), nerve growth factor (NGF), platelet-derived growth factor (PDGF), and insulin-like growth factor (IGF).
  Repetitive high frequency electromagnetic stimulation (rEMS) creates a stimulated focus in the tissue by increasing blood flow and platelets at the capillary level. Electromagnetic stimulation along with growth factors has shown synergetic effects toward enhanced epithelial integrity and neural functions. With the addition of possible iontophoresis effects in the rEMS, the passage of the various active molecules can be augmented at the tissue level thereby increasing the widespread effect of the GFs in the damaged choroidal and outer retinal microenvironment.

SUMMARY:
Purpose: To investigate the efficacy of combined use of retinal repetitive electromagnetic stimulation and subtenon autologous platelet-rich plasma in the treatment of recalcitrant or unresponsive chronic central serous chorioretinopathy.

DETAILED DESCRIPTION:
Central serous chorioretinopathy (CSCR) is a retinal disorder that is mostly unilateral, and predominantly affects young and middle-aged male patients who are otherwise healthy. It is characterized by leaking fluid through a dysfunctional retinal pigment epithelium (RPE) to submacular area resulting in serous neuroretinal detachment. The main risk factors for CSCR include emotional stress, systemic arterial hypertension, pregnancy, use of corticosteroids, and the presence of pachychoroid under the RPE layer.

Although several clinical presentations are described, two forms of CSCR can be distinguished: acute and chronic. Acute CSCR usually presents with sudden visual loss of central vision, disturbed color vision and dark adaptation, central or paracentral scotoma, metamorphopsia, and/or micropsia caused by the rapid accumulation of subretinal fluid (SRF). While spontaneous resolution is common and self-limiting with little or no residual damage in the acute variant, the chronic variant is usually progressive with persistence of SRF. Persistent serous detachment for more than 3 months can result in progressive photoreceptor (PR) compromise, which explains the worsening visual outcomes versus the acute form.

The chronic form of CSCR is characterized by diffuse multifocal irregular hyper-fluorescence seen on fluorescein angiography (FA) and indocyanine green angiography (ICGA) in addition to widespread RPE changes. B-scan optical coherence tompgraphy (OCT) shows elongated PR outer segments and a shallow heterogenous RPE detachment surrounded by subretinal fluid containing fibrin/fluorophore. Widespread diffuse RPE abnormalities including RPE atrophy, intraretinal fluid, and cystic retinal changes, retinal atrophy, subretinal fibrinous accumulation, subretinal fibrosis, and secondary choroidal neovascularization (CNV) are late complications that can lead to permanent visual loss.

The etiology of this disease remains incompletely understood with systemic associations and a complex pathogenesis that involves diffuse dysfunction of the RPE cells, the choroid, or both. Various treatment modalities have been used nowadays with varying success rates. These are selected according to the stage of the disease and diffusiveness and presence of CNV. Examples include acetazolamide, mineralocorticoid receptor antagonists, intravitreal anti-VEGF injections, photodynamic therapy (PDT), and subthreshold micropulse lasers (MPL). However, some of the CSCR cases are recalcitrant or unresponsive to currently available therapy modalities. The disease can be recurrent in 15-50% of cases or bilateral in approximately one-third of cases. Secondary CNV is an important vision-threatening complication of longstanding CSCR with an incidence ranging from 2% to 9%. Thus, new treatment options and approaches, addressing the complex nature of the etiopathogenesis are necessary in patients who would otherwise be disabled.

Platelets are anucleated cells containing many types of growth factors (GFs) such as epithelial growth factor (EGF), fibroblast growth factor (FGF), transforming growth factor (TGF), nerve growth factor (NGF), platelet-derived growth factor (PDGF), and insulin-like growth factor (IGF). These growth factors and their receptors are expressed in epithelial and endothelial cells and play a key role in tissue healing. EGF stimulates the proliferation and migration of epithelial cells. NGF is a neurotrophin that stimulates growth and survival of intraretinal glial cells, Müller's cells, and neurons; it can restore the function of injured neurons. NGF also plays a key role in the integrity and function of the both epithelial cells and nerve fibers. Autologous platelet-rich plasma (aPRP) that contains many GFs has been used to treat retinitis pigmentosa and deep retinal capillary ischemia with promising clinical functional and structural improvements.

Repetitive high frequency electromagnetic stimulation (rEMS) has shown promising potential in epithelization and wound healing. rEMS creates a stimulated focus in the tissue by increasing blood flow and platelets at the capillary level. rEMS can also change the growth factor balance and tyrosine kinase (Trk) receptor activities in damaged microenvironment. Electromagnetic stimulation along with growth factors has shown synergetic effects toward enhanced epithelial integrity and neural functions. With the addition of possible iontophoresis effects in the rEMS, the passage of the various active molecules can be augmented at the tissue level thereby increasing the widespread effect of the GFs in the damaged choroidal and outer retinal microenvironment. Indeed, the combined use of rEMS and aPRP in the treatment of the eyes with deep retinal capillary ischemia due to various etiologies has shown favorable results in otherwise untreatable cases.

The primary aim of this prospective clinical study is to present the utility and efficacy of rEMS together with subtenon aPRP as a new treatment modality in the treatment of chronic CSCR cases which were recalcitrant or unresponsive to the current gold standard treatments. The second aim of the study is to evaluate whether there is ischemic evidences in choriocapillaris and the outer retina as well as their changes with this novel combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* The chronic CSCR cases included here meet one or more of the following criteria:

  * Complaints of recurrent symptoms lasting longer than 3 months;
  * Recalcitrant or unresponsive to all known current treatment modalities including PDT and MPL;
  * Typical B-scan SD-OCT findings of chronicity such as elongation of photoreceptor outer segments indicating chronic nature of sub-macular fluid and/or the presence of serous flat-irregular RPED and focal areas of thickened RPE that lie below the collection of SRF;
  * Widespread RPE/photoreceptor damage, RPE mottling and atrophy along with chronic submacular fluid;
  * Widespread multifocal areas of chronic serous retinal detachment and/or flat-irregular RPEDs in those eyes that effective and reliable laser application is impossible.

Exclusion Criteria:

* Sub-threshold micro-pulse laser and/or photodynamic therapy applied in the last three months;
* Chronic CSCR complicated with secondary CNV.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Sub-macular thickness | Change from baseline sub-macular thickness at 1 months
  This was measured manually from the ellipsoid zone to the Bruch's membrane in where sub-macular fluid is the thickest.

SECONDARY OUTCOMES:
Vessel densities of deep retinal capillary plexus | Change from baseline vessel densities of deep retinal capillary plexus at 1 months
  These were measured with "AngioAnalytic" feature of the OCTA device. To compare the percentage of the vessel densities precisely during follow-up, the "Link-B Scans" button on the screen was activated so that the exact same segmentation planes of the deep capillary plexus could be compared. The OCTA device automatically calculated and displayed the vessel density maps as follow-up sequences (angio retina multi-scan view) and trend analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Umut Arslan, MD, Principal Investigator — Ankara Universitesi Teknokent
Locations (1):
- Ankara University Biotechnology Institute, Ankara, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozmert E, Arslan U. Management of Deep Retinal Capillary Ischemia by Electromagnetic Stimulation and Platelet-Rich Plasma: Preliminary Clinical Results. Adv Ther. 2019 Sep;36(9):2273-2286. doi: 10.1007/s12325-019-01040-2. Epub 2019 Aug 5. PMID 31385285
- [Result] Nicholson B, Noble J, Forooghian F, Meyerle C. Central serous chorioretinopathy: update on pathophysiology and treatment. Surv Ophthalmol. 2013 Mar-Apr;58(2):103-26. doi: 10.1016/j.survophthal.2012.07.004. PMID 23410821
- [Result] Manayath GJ, Ranjan R, Karandikar SS, Shah VS, Saravanan VR, Narendran V. Central serous chorioretinopathy: Current update on management. Oman J Ophthalmol. 2018 Sep-Dec;11(3):200-206. doi: 10.4103/ojo.OJO_29_2018. PMID 30505108
- [Result] Ross A, Ross AH, Mohamed Q. Review and update of central serous chorioretinopathy. Curr Opin Ophthalmol. 2011 May;22(3):166-73. doi: 10.1097/ICU.0b013e3283459826. PMID 21427570
- [Result] Gemenetzi M, De Salvo G, Lotery AJ. Central serous chorioretinopathy: an update on pathogenesis and treatment. Eye (Lond). 2010 Dec;24(12):1743-56. doi: 10.1038/eye.2010.130. Epub 2010 Oct 8. PMID 20930852
- [Result] Arslan U, Ozmert E, Demirel S, Ornek F, Sermet F. Effects of subtenon-injected autologous platelet-rich plasma on visual functions in eyes with retinitis pigmentosa: preliminary clinical results. Graefes Arch Clin Exp Ophthalmol. 2018 May;256(5):893-908. doi: 10.1007/s00417-018-3953-5. Epub 2018 Mar 15. PMID 29546474
- [Derived] Arslan U, Ozmert E. Treatment of resistant chronic central serous chorioretinopathy via platelet-rich plasma with electromagnetic stimulation. Regen Med. 2020 Aug;15(8):2001-2014. doi: 10.2217/rme-2020-0056. Epub 2020 Oct 27. PMID 33107400